CLINICAL TRIAL: NCT04060225
Title: Short-term and Intermediate-term Effects of High Volume High Caffeine Content Coffee on Blood Pressure in Young Adults
Brief Title: Effects of High Caffeine Content Coffee on Blood Pressure in Young Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not possible to enroll during COVID pandemic
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, John Bisognano, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00003172
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants will be asked to participate in a single arm study with three phases (washout phase, abstinence phase, and exposure phase). These participants will first be asked to abstain from drinking any caffeinated food or beverages for 72 hours (known as the washout phase). Following the first phase, participants will then wear a blood pressure cuff to collect diastolic and systolic blood pressure for 24 hours (abstinence phase) wherein they will be asked to refrain from caffeinated products. Participants will then drink the coffee intervention and collect blood pressure measurements for 24 hours (exposure phase).
  Interventions: Other: Coffee

INTERVENTIONS:
Other: Coffee — Starbuck's brand blonde roast coffee, 20 ounces

SUMMARY:
The purpose of this study is to help further the understanding of the effects of commercially available high-caffeine containing coffee on blood pressure in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Male or Female
* No prior diagnosis of hypertension
* No prior chronic disease requiring medical intervention
* Ability to demonstrate correct usage of ambulatory blood pressure monitoring device

Exclusion Criteria:

- Age less than 18 years old

* Prior chronic disease (such as hypertension) requiring medical intervention
* Previously undiagnosed hypertension
* Intolerance or allergy to coffee or caffeine
* Inability to demonstrate correct usage of ambulatory blood pressure monitoring device
* Inability to complete the required abstinence period prior to study interventions
* Known pregnancy
* Use of birth control
* Tobacco use
* Participation in other investigational drug studies at the time of this study
* Medical illness requiring medical or symptomatic management

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Mean change ambulatory blood pressure | baseline to 30 minutes
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 0-3 hour after drinking the coffee versus 0-3 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 1 hour
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 0-3 hour after drinking the coffee versus 0-3 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 1.5 hour
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 0-3 hour after drinking the coffee versus 0-3 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 2 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 0-3 hours after drinking the coffee versus 0-3 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 2.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 0-3 hours after drinking the coffee versus 0-3 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 3 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 0-3 hour after drinking the coffee versus 0-3 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 3.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 3-6 hours after drinking the coffee versus 3-6 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 4 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 3-6 hours after drinking the coffee versus 3-6 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 4.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 3-6 hours after drinking the coffee versus 3-6 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 3-6 hours after drinking the coffee versus 3-6 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 5.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 3-6 hours after drinking the coffee versus 3-6 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 6 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 3-6 hours after drinking the coffee versus 3-6 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 6.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 6-9 hours after drinking the coffee versus 6-9 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 7 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 6-9 hours after drinking the coffee versus 6-9 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 7.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 6-9 hours after drinking the coffee versus 6-9 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 8 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 6-9 hours after drinking the coffee versus 6-9 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 8.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 6-9 hours after drinking the coffee versus 6-9 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 9 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 6-9 hours after drinking the coffee versus 6-9 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 9.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 9-12 hours after drinking the coffee versus 9-12 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 10 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 9-12 hours after drinking the coffee versus 9-12 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 10.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 9-12 hours after drinking the coffee versus 9-12 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 11 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 9-12 hours after drinking the coffee versus 9-12 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 11.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 9-12 hours after drinking the coffee versus 9-12 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 12 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 9-12 hours after drinking the coffee versus 9-12 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 12.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 12-15 hours after drinking the coffee versus 12-15 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 13 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 12-15 hours after drinking the coffee versus 12-15 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 13.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 12-15 hours after drinking the coffee versus 12-15 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 14 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 12-15 hours after drinking the coffee versus 12-15 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 14.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 12-15 hours after drinking the coffee versus 12-15 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 15 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 12-15 hours after drinking the coffee versus 12-15 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 15.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 15-18 hours after drinking the coffee versus 15-18 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 16 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 15-18 hours after drinking the coffee versus 15-18 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 16.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 15-18 hours after drinking the coffee versus 15-18 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 17 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 15-18 hours after drinking the coffee versus 15-18 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 17.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 15-18 hours after drinking the coffee versus 15-18 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 18 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 15-18 hours after drinking the coffee versus 15-18 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 18.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 18-21 hours after drinking the coffee versus 18-21 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 19 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 18-21 hours after drinking the coffee versus 18-21 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 19.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 18-21 hours after drinking the coffee versus 18-21 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 20 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 18-21 hours after drinking the coffee versus 18-21 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 20.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 18-21 hours after drinking the coffee versus 18-21 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 21 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 18-21 hours after drinking the coffee versus 18-21 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 21.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 21-24 hours after drinking the coffee versus 21-24 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 22 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 21-24 hours after drinking the coffee versus 21-24 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 22.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 21-24 hours after drinking the coffee versus 21-24 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 23 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 21-24 hours after drinking the coffee versus 21-24 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 23.5 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 21-24 hours after drinking the coffee versus 21-24 hours after the end of the washout period.
Mean change ambulatory blood pressure | baseline, 24 hours
  Participants will wear a ambulatory blood pressure cuff for 24 hours with half hourly measurements of systolic and diastolic blood pressure. Mean change will be measured comparing the same participants blood pressure at 21-24 hours after drinking the coffee versus 21-24 hours after the end of the washout period.

CONTACTS AND LOCATIONS:
Locations (1):
- URMC Cardiology; 919 Westfall Rd, Building C, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No